CLINICAL TRIAL: NCT03994068
Title: VIVO Non-invasive Time Assessment Protocol
Brief Title: VIVO Mapping Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VIVO-RBH01
Record Dates: First submitted 2019-05-04; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Ventricular Tachycardia; Ventricular Ectopic Beat(S)
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VIVO mapping pre-procedure (Experimental): 15 patients with structurally normal heart and indication for PVC/VT catheter ablation, who will undergo pre-procedural non invasive mapping with VIVO mapping system.
  Interventions: Diagnostic Test: VIVO non invasive mapping

INTERVENTIONS:
Diagnostic Test: VIVO non invasive mapping — non invasive pre-procedural localization of PVC / VT origin

SUMMARY:
This is a single centre study enrolling 15 subjects with structurally normal hearts that are already indicated for a ventricular ablation procedure (VT or PVCs).

The purpose is to compare the accuracy of VIVO and to assess its efficacy to decrease procedural time, and ideally, the procedural overall costs, as compared to standard of care ablation procedures. Results will be compared with data from

DETAILED DESCRIPTION:
VIVO TM is a non invasive mapping system which can be used to localize PVC / VT origin prior to the ablative procedure.

Subjects scheduled for catheter ablation with VIVO will undergo a CT scan prior to the procedure, which will be used to create a personalized 3D model. This will be merged with a 3D photograph (taken at the start of the procedure) of the ECG electrodes on the subject's torso.

Then, the recording of the 12 lead ECG will be imported into the VIVO software. All of this data will be combined via the software and a mathematical algorithm will determine the origin of the arrhythmia. This will show the physician where to perform a successful ablation. After 3 months, the subject will return for follow up and will receive another ECG Holter monitor (ECG recording) to determine ablation success.

Subjects will be exited from the study after the 3 month follow up visit. Patients will receive standard clinical care prior to, during and after their scheduled procedure, as well as after being discarded from the trial.

Results will be analysed and compared to those from an historical cohort of patients (age / gender matched, undergone the same procedure) ablated by the same operator within the previous 5 years (from a database already collected). Data will be anonymised as per current regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are at least 18 years or older
2. Subjects who are scheduled for PVC/VT ablation procedure
3. Subjects who have signed an IRB/EC approved Informed Consent Form and applicable subject privacy protection authorization per local law
4. Subjects will be selected without regard to gender or age (unless precluded by local regulatory requirements)
5. Subjects with or without cardiac structural disease

Exclusion Criteria:

1. Reversible causes of PVC/VT
2. Subjects with recent (within 3 months) acute coronary syndrome
3. Subjects who are contraindicated for CT or MRI (must be able to get one)
4. Subject whose MRI or CT scan does not comply with the requirements of this protocol
5. Subjects who are contraindicated for an electrophysiology procedure and/or fluoroscopy:

   * INR > 3.5
   * Active infection
   * Pregnancy: Females of childbearing potential with a positive pregnancy test.
6. Existing mechanical heart valve
7. Subjects with structural cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of procedural time (in minutes) | three months
  Use of VIVO mapping to localize the PVC / VT origin prior to the catheter procedure in order to change procedural time. Procedural time is meant to be measured in minutes per procedure, and it is normally considered from "puncture time" to "sheaths removal".
Safety - absence of acute adverse events using VIVO system for non-invasive mapping | three months
  Absence of acute adverse events due to the use of VIVO system during PVC/VT ablation in the cohort of patients enrolled for the study. Acute adverse events are described in section 12 of the study protocol and will be reported in specific forms to the Sponsor and REC.
Safety 2 - absence of acute adverse events using VIVO system for mapping and during the whole ablation procedure | three months
  Safety endpoint of the entire mapping and ablation strategy, determined by the absence of adverse events (AEs).

SECONDARY OUTCOMES:
economical outcome: change of procedural costs | three months
  To assess economical outcome, which is meant as cost change (in pounds) per number of cases
clinical outcome assessed as change of PVCs/VT burden | three months
  Count of PVC/VT burden at 3-month follow up Holter (expressed as No. / 24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Ernst, MD, PhD, Principal Investigator — Royal Brompton and Harefield Hospital Trust; Ilaria Cazzoli, MD, Study Chair — Royal Brompton and Harefield Hospital Trust

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT03994068/Prot_SAP_000.pdf